CLINICAL TRIAL: NCT05369351
Title: Efficacy and Safety of Mirabegron in Intracerebral Hemorrhage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Liu, Professor of Neurology Department, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2022-YX-073-01
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment+mirabegron (Experimental): In addition to standard treatment, the first dose of mirabegron 50mg/day will be given within 72 hours of symptom onset and continued until the 7th day after onset.
  Interventions: Drug: Standard treatment+mirabegron
- Standard treatment (Other): Patients will receive usual care
  Interventions: Other: Standard treatment

INTERVENTIONS:
Drug: Standard treatment+mirabegron — In addition to standard treatment, the first dose of mirabegron 50mg/day will be given within 72 hours of symptom onset and continued until the 7th day after onset.
  Arms: Standard treatment+mirabegron
Other: Standard treatment — Standard treatment
  Arms: Standard treatment

SUMMARY:
Intracerebral hemorrhage (ICH) accounts for 10-15% of all strokes without effective pharmacological treatment. Inflammation following ICH contributes to barrier disruption and peri-hematoma edema, leading to deterioration of neurological function. Preclinical evidence suggests that bone marrow hematopoietic stem and progenitor cells (HSPCs) are swiftly activated after ICH. Thereafter, these HSPCs produce an increased output of anti-inflammatory monocytes as an endogenous protective mechanism. Stimulation of β3 adrenergic receptor using selective agonists promotes the production of anti-inflammatory monocytes in bone marrow, and thereby reduces neuroinflammation, brain edema and neurological deficits. This study is to assess the safety and efficacy of a β3 adrenergic receptor agonist Mirabegron as a potential treatment option in ICH patients.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy and safety of mirabegron in patients with intracerebral hemorrhage based on standard therapy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged above 18 years old.
2. The volume of the hematoma is 5-30 ml (including the cerebral cortex; Putamen, thalamus, caudate nucleus and related deep tracts; Cerebellar hemorrhage), which determined by CT scan.
3. The onset of cerebral hemorrhage symptoms or the time from last normal to detection is not more than 72 hours.
4. Patients with Glasgow Coma Scale (GCS) score ≥6 and < 12.
5. Before the onset of the disease, function was independent and mRS score<1.
6. Able and willing to sign written informed consent and comply with the requirements of the research protocol.

Exclusion criteria:

1. Multifocal cerebral hemorrhage, brain stem hemorrhage, or ventricular hemorrhage.
2. Secondary cerebral hemorrhage caused by aneurysm, brain tumor, arteriovenous malformation, thrombocytopenia, coagulation disorder, traumatic brain injury, etc.
3. Patients who require hematoma removal surgery or other emergency surgical interventions (such as decompressive craniectomy), or who are critically ill and close to death.
4. Patients who interfere with drug use due to nausea or vomiting.
5. Combined with the following conditions that preclude participation in the study due to other systemic diseases: Severe hepatic or renal impairment, atrial fibrillation or tachycardia, pulmonary infection, severe urinary tract infection, severe urinary tract obstruction, medically uncontrolled hypertension (systolic blood pressure ≥180mmHg or diastolic blood pressure ≥110mmHg), pregnant and lactating women, and a history of malignant tumors within 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Changes in absolute perihematomal edema volume measured by computed tomography (CT) | 7 and 14 days
  Repeated CT images will be obtained at 24-48 hours after diagnosis and on days 7 and 14 with CT at 24-48 hours after diagnosis as the baseline for analysis.

SECONDARY OUTCOMES:
Changes in absolute hematoma volume measured by CT after ICH | 7 and 14 days
  Repeated CT images will be obtained at 24-48 hours after diagnosis and on days 7 and 14 with CT at 24-48 hours after diagnosis as the baseline for analysis.
Changes in NIHSS scores | 7 and 14 days
  The assessment will be based on the National Institutes of Health Stroke Scale (NIHSS) with a score range of 0 (asymptomatic) to 42 (death).
The rate of functional independence at 90 days | 90 days
  Number of participants with functional independence. Modified Rankin scale (mRS) is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes neurological disability.
  Functional Independence:
  0 - no symptoms at all
  1 - no significant disability despite symptoms; able to carry out all usual duties and activities 2- slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
Proportion of adverse drug reactions | 14 days
  Adverse events related to mirabegron will be recorded.
All cause mortality | 90 days
  Death induced by any cause
Changes of immune cells in peripheral blood | 14 days
  The counts of monocytes subsets and other immune cells in peripheral blood were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China